CLINICAL TRIAL: NCT00572962
Title: Prospective Clinical Observational Cohort Study to Evaluate the Use of a Tissue Separating Mesh (Proceed®) in Laparoscopic Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/268
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): use of a tissue separating mesh (Proceed®) in Laparoscopic Ventral hernia repair
  Interventions: Procedure: use of a tissue separating mesh (Proceed®) in Laparoscopic Ventral hernia repair

INTERVENTIONS:
Procedure: use of a tissue separating mesh (Proceed®) in Laparoscopic Ventral hernia repair — use of a tissue separating mesh (Proceed®) in Laparoscopic Ventral hernia repair

SUMMARY:
1. General: antibiotic prophylaxis: cefazoline (Cefacidal™) 2 gram iv administered 30 minutes before surgery
2. Laparoscopic surgery

   * at least 5 cm overlap (mesh diameter should exceed hernia size by at least 10 cm)
   * with or without anchoring transparietal sutures or double crown technique

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from the patient or his/her legal representative
* ventral hernia requiring elective surgical repair

Exclusion Criteria:

* no written informed consent
* 'hostile' abdomen; open abdomen treatment
* contraindication to pneumoperitoneum
* emergency surgery (incarcerated hernia)
* parastomal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
recurrence rate | after 1 year

SECONDARY OUTCOMES:
morbidity rate | perioperative
quality of life | after 1 year
postoperative pain | within 1 week
long term complication rate | after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Berrevoet F, Tollens T, Berwouts L, Bertrand C, Muysoms F, De Gols J, Meir E, De Backer A. A belgian multicenter prospective observational cohort study shows safe and efficient use of a composite mesh with incorporated oxidized regenerated cellulose in laparoscopic ventral hernia repair. Acta Chir Belg. 2014 Jul-Aug;114(4):233-8. PMID 26021417
- See also: Website University Hospital Ghent — http://www.uzgent.be